CLINICAL TRIAL: NCT02084485
Title: A Randomized, Double-blind, Placebo-controlled, 2-way Crossover Study to Determine the Effects of a Single Oral Dose of Ph-797804 on Induced Sputum Inflammatory Markers Following Inhaled Lipopolysaccharide (Lps) Challenge in Healthy Volunteers
Brief Title: PH-797804 LPS Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: A6631010
Record Dates: First submitted 2014-03-03; First posted 2014-03-12 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: COPD; LPS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — PH 797804

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: PH-797804
- Arm B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PH-797804 — 30 MG Single dose
  Arms: Arm A
Drug: Placebo — matching placebo
  Arms: Arm B

SUMMARY:
The study was performed to assess the effect of PH-797804 on neutrophils (white cells) in the sputum after a challenge with an endotoxin (inhaled LPS). Neutrophils are a sign of inflammation and PH-797804 is being developed as a potential anti-inflammatory treatment for patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female (WONCBP), non atopic volunteers aged 18-50 years
* Able to produce sputum

Exclusion Criteria:

* Current Smokers
* Abnormal liver function test
* Respiratory Tract Infection within 4 weeks

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Sputum Cell Counts | 6 hours post LPS challenge
  Neutrophil & Macrophage count (total and differential)
Sputum Cytokines | 6 hours post LPS challenge
  TNF-α, MIP-1β, IL-6, MPO, MCP-1, GRO-α

SECONDARY OUTCOMES:
Systemic Inflammatory Indices | 1, 4, 6 and 7 hours post LPS
  Neutrophil count, GRO-α, TNF-α, MIP-1β, IL-6, MPO, MCP-1, CRP

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Denmark Hill, London, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631010&StudyName=PH-797804%20LPS%20study%20in%20Healthy%20Volunteers